CLINICAL TRIAL: NCT02534025
Title: Remote Ischemic Preconditioning in Liver Transplantation
Acronym: RIRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1/2015
Record Dates: First submitted 2015-08-09; First posted 2015-08-27 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Liver Transplanatation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- P group (Experimental): Elevation of Cuff pressure to 200 mm Hg for 5 minutes four times 5 minutes apart
  Interventions: Procedure: Ischemia preconditioining
- C group (No Intervention): no intervention will be added to routine anesthetic mangement

INTERVENTIONS:
Procedure: Ischemia preconditioining — Elavate blood pressure cuff pressure to 200
  Arms: P group

SUMMARY:
Remote (upper arm) ischemic preconditioning in the donor of living donor liver transplanta to ameliorate the effect of reperfusion injury in recipients.

DETAILED DESCRIPTION:
Upper arm ischemia will be induced by elevation of NIBP cuff pressure to 200 mm Hg for 5 minutes repeated four times 5 mniutes apart, aiming to decrease the effect of ischemia reperfusion in the graft liver.

ELIGIBILITY:
Inclusion Criteria:

* All candidates for living donor liver transplantation

Exclusion Criteria:

* Donors with peripheral vascular disease

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
liver enzymes ( SGOT and SGPT) as indicator of graft injury | 30 minutes
  Hemodynamic effects of reperfusion ijury

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dkahleya, Egypt